CLINICAL TRIAL: NCT06032585
Title: TRANSPARK_LONG: The Diagnostic Value of Early Transcranial Ultrasound in Patients With Extrapyramidal Diseases in a Swedish Population: an Evaluation in the Form of a Retrospective Cohort Study With a Long Follow-up Time
Brief Title: TRANSPARK_LONG: The Diagnostic Value of Early Transcranial Ultrasound in Patients With Extrapyramidal Diseases in a Swedish Population
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: Dnr 2022-06697-01
Record Dates: First submitted 2023-09-04; First posted 2023-09-13 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Parkinsonism; Tremor; Dementia
Keywords: Transcranial ultrasound; Substantia nigra
MeSH Terms: conditions — Parkinsonian Disorders; Tremor; Dementia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with parkinsonism: Parkinsonism incl. tremor, parkinsons, atypical parkinsons

SUMMARY:
Popular science summary of the project The purpose of the study is to investigate in a Swedish population how well the investigators' previous ultrasound findings match the final diagnosis (PD, APS or ET) after a particularly long follow-up time, which greatly increases the certainty that the diagnosis does not change more and is thus correct. Furthermore, the investigators want to study whether the initial ultrasound findings have changed during the control interval and whether measurement results regarding the diameter in one of the fluid-filled rooms in the brain (third ventricle) can be correlated with the development of cognitive impairment or dementia later in the course of the disease. For this, this study have got ethical permission to go into the patients' medical records and to call a subgroup back to the clinic to be able to do a new examination and a memory test.

ELIGIBILITY:
Inclusion Criteria:

* Patients with parkinsonism or essential tremor who came into contact with our clinic before 2017
* Satisfactory transcranial bone window
* Previous TU (clinical indication)

Exclusion Criteria:

* No transcranial bone window

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosted patients with parkinsonism between 2013-2017 at our centre
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Correlation | over 7-10 yrs
  Is hyperechogenicity of substantia nigra at mesencephal plane (measured bilaterally in mm2 by transcranial b-mode sonography correlated with a high percentage of patients with classical Parkinsons Disease in contrast to atypical parkinsonism patients?

SECONDARY OUTCOMES:
Correlation | 7-10 (retrospective)
  Is 3rd ventricle atrophy (measured in mm by b-mode transcranial sonography) correlated with a high % of demented patients in the cohort?

CONTACTS AND LOCATIONS:
Locations (1):
- Skåne Univ Hospital, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided